CLINICAL TRIAL: NCT03934710
Title: Mood Effects of Serotonin Agonists Extended
Acronym: MESA-E
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB18-1183; 5R01DA002812 (NIH)
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — Serotonin Receptor Agonists; Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Serotonin agonist 13ug (Experimental): 13ug of serotonin agonist
  Interventions: Drug: Serotonin agonist - 13ug
- Serotonin agonist 26ug (Experimental): 26ug of serotonin agonist
  Interventions: Drug: Serotonin agonist - 26ug

INTERVENTIONS:
Drug: Placebo — Drug will be administered in solution form
  Arms: Placebo
Drug: Serotonin agonist - 13ug — 13ug lysergic acid diethylamide
  Other Names: LSD
  Arms: Serotonin agonist 13ug
Drug: Serotonin agonist - 26ug — 26ug lysergic acid diethylamide
  Other Names: LSD
  Arms: Serotonin agonist 26ug

SUMMARY:
In this study we are examining the effects of repeated very low doses of serotonin agonists on mood individuals with negative mood.

DETAILED DESCRIPTION:
Here, we are examining the effects of four repeated low doses of lysergic acid diethylamide (LSD), compared to placebo, administered to healthy adults at 3-4 day intervals, on mood, cognitive performance and responses to emotional tasks

ELIGIBILITY:
Inclusion Criteria:

* English fluency
* High school level education
* BMI between 19 and 30

Exclusion Criteria:

* Diagnosed medical condition
* women who are nursing, pregnant, or plan to become pregnant within 3 months
* History of psychotic disorder or family history of psychotic disorder

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, Principal Investigator — University of Chicago
Locations (1):
- Matthew Bona, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Serotonin Agonist: 13ug of serotonin agonist
  Serotonin agonist: 13ug lysergic acid diethylamide
- Serotonin Agonist: 26ug of serotonin agonist: 26ug lysergic acid diethylamide
Period: Overall Study
Arm/Group | Placebo | Serotonin Agonist | Serotonin Agonist
Started | 18 | 19 | 19
Completed | 18 | 19 | 19
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Serotonin Agonist 13ug: 13ug of serotonin agonist
  Serotonin agonist: 13ug lysergic acid diethylamide
- Serotonin Agonist 26 ug: 26ug of serotonin agonist
  Serotonin agonist: 26ug lysergic acid diethylamide
- Total: Total of all reporting groups
Arm/Group | Placebo | Serotonin Agonist 13ug | Serotonin Agonist 26 ug | Total
Number analyzed (Participants) | 18 | 19 | 19 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 19 | 56
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 6 | 19
  Male | 11 | 13 | 13 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 12 | 11 | 13 | 36
  More than one race | 5 | 4 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 19 | 56
Education - High School Education [Count of Participants; unit: Participants] | 18 | 19 | 19 | 56

OUTCOME MEASURES:

1. Primary Outcome: DASS-21
Description: The primary outcome measure is the depression anxiety and stress scale (DASS) 21. This self-report measure contains 21 items and the range of scores for depression is 0-42, anxiety 0-42, and stress 0-42. Our primary outcome measure is total depression scale ratings during session 5, with lower scores indicating lower ratings of depression.
Time Frame: End of session 5, approximately 2 weeks from baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Serotonin Agonist 26ug: Serotonin agonist: 26 ug lysergic acid diethyl amide
Arm/Group | Placebo | Serotonin Agonist 13ug | Serotonin Agonist 26ug
Number analyzed (Participants) | 18 | 19 | 19
units on a scale | 2.9 (3) | 2.7 (2.9) | 4.5 (3.7)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 weeks.
Groups:
- Serotonin Agonist 13 ug: 13ug of serotonin agonist
  Serotonin agonist: 13ug lysergic acid diethylamide
Arm/Group | Placebo | Serotonin Agonist 13 ug | Serotonin Agonist 26 ug
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03934710/Prot_SAP_000.pdf